CLINICAL TRIAL: NCT00019630
Title: Phase I Study of Doxorubicin HCl Liposome in Pediatric Patients With Refractory Solid Tumors
Brief Title: Liposomal Doxorubicin in Treating Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066924; NCI-99-C-0039F; LIPO-NCI-99-C-0039; NCI-99-C-0039; NCT00001798 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Childhood Soft Tissue Sarcoma; Childhood Liver Cancer; Bone Cancer; Brain Tumor; Kidney Tumor
Keywords: Ewing's family of tumors; Wilms' tumor; adult solid tumor; body system/site cancer; bone cancer; brain tumor; cancer; central nervous system cancer; childhood brain stem glioma; childhood brain tumor; childhood cancer; childhood central nervous system germ cell tumor; childhood cerebellar astrocytoma; childhood cerebral astrocytoma; childhood choroid plexus tumor; childhood craniopharyngioma; childhood ependymoma; childhood extracranial germ cell tumor; childhood extragonadal malignant germ cell tumor; childhood liver cancer; childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; childhood mature and immature teratomas; childhood medulloblastoma; childhood meningioma; childhood oligodendroglioma; childhood rhabdomyosarcoma; childhood soft tissue sarcoma; childhood solid tumor; childhood supratentorial primitive neuroectodermal and pineal tumors; childhood visual pathway and hypothalamic glioma; endocrine cancer; gastrointestinal cancer; genetic condition; kidney tumor; kidney/urinary cancer; liver and intrahepatic biliary tract cancer; muscle cancer; musculoskeletal cancer; neuroblastoma; osteosarcoma; osteosarcoma/malignant fibrous histiocytoma of bone; pediatric germ cell tumor; previously treated childhood rhabdomyosarcoma; recurrent Wilms' tumor; recurrent childhood brain stem glioma; recurrent childhood brain tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood liver cancer; recurrent childhood malignant germ cell tumor; recurrent childhood medulloblastoma; recurrent childhood rhabdomyosarcoma; recurrent childhood soft tissue sarcoma; recurrent childhood supratentorial primitive neuroectodermal and pineal tumors; recurrent childhood visual pathway and hypothalamic glioma; recurrent neuroblastoma; recurrent osteosarcoma; recurrent tumors of the Ewing's family; solid tumor; stage, Ewing's family of tumors; stage, Wilms' tumor; stage, childhood extracranial germ cell tumor; stage, childhood liver cancer; stage, childhood medulloblastoma; stage, childhood rhabdomyosarcoma; stage, childhood soft tissue sarcoma; stage, neuroblastoma; stage, osteosarcoma; stage/type, childhood brain tumor; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Bone Neoplasms; Brain Neoplasms; Carcinoma, Renal Cell; Neuroectodermal Tumors, Primitive, Peripheral; Wilms Tumor; Neoplasms; Central Nervous System Neoplasms; Astrocytoma; Choroid Plexus Neoplasms; Familial ependymoma; Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma; Medulloblastoma; Meningioma; Oligodendroglioma; Pinealoma; Optic Nerve Glioma; Endocrine Gland Neoplasms; Gastrointestinal Neoplasms; Genetic Diseases, Inborn; Urologic Neoplasms; Carcinoma, Hepatocellular; Muscle Neoplasms; Neuroblastoma; Osteosarcoma; Histiocytoma, Malignant Fibrous

INTERVENTIONS:
Drug: doxorubicin HCl liposome

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of liposomal doxorubicin in treating children who have refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the tolerance to and toxicity profile of doxorubicin HCl liposome (Lipodox) at standard doxorubicin doses and doses of Lipodox that were tolerable in adults administered every 3 weeks in pediatric patients with refractory solid tumors.

II. Determine the maximum tolerated dose of this drug in these patients if dose-limiting toxicity is observed at doses of 105 mg/m2 or less.

III. Determine the pharmacokinetics of this drug in these patients. IV. Assess the cardiotoxicity of this drug in children who have previously been treated with free doxorubicin and in children who have not previously received doxorubicin.

V. Evaluate the feasibility of using cardiac MRI functional imaging as a screening tool for the quantitative assessment of doxorubicin-induced cardiotoxicity.

VI. Determine if serum troponin t levels are a useful biomarker for doxorubicin-induced myocardial damage.

PROTOCOL OUTLINE: This is a dose-escalation, multicenter study. Patients receive doxorubicin HCl liposome IV over 60 minutes. Treatment repeats every 4 weeks for a maximum of 10 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 4-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 4 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL:

A total of 21-36 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically confirmed solid tumor, including but not limited to: Rhabdomyosarcoma and other soft tissue sarcomas Ewing's family tumors Osteosarcoma Neuroblastoma Wilms' tumor Hepatic tumors Germ cell tumors Primary brain tumors Histological confirmation for brain stem gliomas may be waived Refractory to standard treatment and no curative therapy available Measurable or evaluable disease Evidence of progressive disease on prior chemotherapy or radiotherapy or persistent disease after prior surgery --Prior/Concurrent Therapy-- Biologic therapy: At least 1 week since prior colony-stimulating factors (e.g., filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa) At least 4 months since prior bone marrow transplantation No concurrent anticancer immunotherapy Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy (4 weeks for nitrosoureas) and recovered Prior anthracyclines as adjuvant front-line therapy allowed provided: No relapse during therapy At least 6 months since last dose Cumulative dose is no greater than 400 mg/m2 for patients who received bolus administration without a concurrent cardioprotectant (e.g., dexrazoxane) or received cardiac irradiation and no greater than 450 mg/m2 for patients who received either continuous infusion or administration with a concurrent cardioprotectant and have not received cardiac irradiation No other concurrent anticancer chemotherapy Endocrine therapy: Concurrent corticosteroids for brain tumor-associated edema allowed (must be on stable or decreasing dose for at least 1 week prior to study) Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No more than 1,500 cGy of prior cardiac radiotherapy No prior extensive radiotherapy (e.g., craniospinal radiation, total body radiation, or radiation to more than half of the pelvis) No concurrent anticancer radiotherapy Surgery: See Disease Characteristics Other: No other concurrent anticancer investigational agents No other concurrent liposomal formulations of any drug (e.g., liposomal amphotericin B) --Patient Characteristics-- Age: 21 and under Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: Absolute granulocyte count greater than 1,500/mm3 Hemoglobin greater than 8 g/dL Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGPT no greater than 2 times upper limit of normal No significant hepatic dysfunction Renal: Creatinine normal OR Creatinine clearance at least 60 mL/min Cardiovascular: Cardiac ejection fraction at least 45% on MUGA (National Cancer Institute patients) OR Shortening fraction at least 28% on echocardiogram (Children's Hospital of Philadelphia patients) No significant or preexisting cardiac dysfunction (e.g., recurrent or persistent cardiac dysrhythmia or an ejection fraction below the lower limit of normal on MUGA or echocardiogram) Pulmonary: No significant pulmonary dysfunction Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No clinically significant unrelated systemic illness (e.g., serious infections or organ dysfunction) No allergy to doxorubicin or other anthracyclines, eggs, egg products, or other liposomal drug formulations

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lowe, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Pediatric Oncology Branch, Bethesda, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania